CLINICAL TRIAL: NCT07279688
Title: Justification And Evaluation of Baricitinib Plus Corticosteroids Versus corticosteroiDs Alone in pOlymyalgia RhEumatica - JADORE-BARI Study
Brief Title: Justification And Evaluation of Baricitinib Plus Corticosteroids Versus corticosteroiDs Alone in pOlymyalgia RhEumatica
Acronym: JADORE-BARI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 29BRC23.0160 - JADORE-BARI
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Polymyalgia Rheumatica (PMR)
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — baricitinib; Tablets

STUDY DESIGN:
Intervention Model Description: This is a multicentre double blinded randomized (1:1:1 ratio) placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 4 mg (Active Comparator): Oral baricitinib 4 mg for 12 weeks; Oral GCs prescribed at baseline Then, at week 12, if PMR-AS ≤10, patients will receive baricitinib 4 mg for 12 weeks. If PMR-AS >10, they will receive GCs according to the PMR-AS. Dosage of GCs will be decreased (1 mg every week) or increased according to PMR-AS (PMR-AS <10: decrease, PMR-AS >20 increase, 10≤ PMR-AS ≤20: stable dose) according to investigator's opinion.
  Interventions: Drug: Baricitinib 4 MG Oral Tablet; Drug: Placebo 2 mg
- Experimental group 2 mg (Active Comparator): Oral baricitinib 2 mg for 12 weeks; Oral GCs prescribed at inclusion Then, at week 12, if PMR-AS ≤10, patients will receive baricitinib 2 mg for 12 weeks. If PMR-AS >10, they will receive GCs according to the PMR-AS. Dosage of GCs will be decreased (1 mg every week) or increased according to PMR-AS (PMR-AS <10: decrease, PMR-AS >20 increase, 10≤ PMR-AS ≤20: stable dose) according to investigator's opinion.
  Interventions: Drug: Baricitinib 2 MG Oral Tablet; Drug: Placebo 4 mg
- Control group (Placebo Comparator): Oral placebo for 12 weeks; Oral GCs at inclusion. Then, at week 12, if PMR-AS ≤10, placebo for 12 weeks. If PMR-AS >10, they will receive GCs according to the PMR-AS. Dosage of GCs will be decreased (1 mg every week) or increased according to PMR-AS (PMR-AS <10: decrease, PMR-AS >20: increase, 10≤ PMR-AS ≤20: stable dose) and according to investigator's opinion.
  Interventions: Drug: Placebo 4 mg; Drug: Placebo 2 mg

INTERVENTIONS:
Drug: Baricitinib 4 MG Oral Tablet — Patient will take a tablet of 4 mg/d during 12 weeks and then 4 mg/d during 12 weeks if the patient achieves PMR-AS≤ 10 at week 12.
  Arms: Experimental group 4 mg
Drug: Baricitinib 2 MG Oral Tablet — Patient will take a tablet of 2 mg/d during 12 weeks and then 2 mg/d during 12 weeks if the patient achieves PMR-AS≤ 10 at week 12.
  Arms: Experimental group 2 mg
Drug: Placebo 4 mg — Patient will take a tablet of placebo for 12 weeks and then placebo during 12 weeks if the patient achieves PMR-AS ≤ 10 at week 12.
  Arms: Control group; Experimental group 2 mg
Drug: Placebo 2 mg — Patient will take a tablet of placebo for 12 weeks and then placebo during 12 weeks if the patient achieves PMR-AS ≤ 10 at week 12.
  Arms: Control group; Experimental group 4 mg

SUMMARY:
Polymyalgia rheumatic (PMR) is an inflammatory rheumatic disease affecting the elderly. The diagnosis is based on established ACR/EULAR classification criteria.

The activity of the disease is evaluated using the PMR-AS, a disease activity score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment and pain assessment measured by the patient using VAS, and the C-reactive protein (CRP) level. The PMR-AS-CRP (PMR-AS) is considered as relevant to define disease activity (low activity <7; moderate activity 7 to 17; high activity >17), flare (>10), remission (<1.5), but also to decide if treatment has to be decreased, unchanged or increased (PMR-AS <10: decrease, PMR-AS >20 increase, 10≤ PMR-AS ≤20: stable dose) [10-12].

Long term low-dose glucocorticoid (GCs) (prednisone or prednisolone started at 12.5 to 25 mg/day progressively tapered) is the mainstay of the treatment. But comorbidities in PMR are due to GCs and 30% of the patients underwent a relapse when tapering GCs.

Today, the physicians do not know what is the best duration and the best dosage of GCs. The international recommendation suggests to start prednisone at a dose between 12.5 to 25 mg, to be at 10 mg at 1 or 2 months, and then to decrease slowly. The treatment is generally ordered for 6-18 months but it is possible to try a shorter treatment duration when patients have been previously treated with GCs or in case of comorbidities.

The TENOR study, a phase 2 study, demonstrated efficacy of tocilizumab as first line treatment in PMR and its ability to spare GCs. The Semaphore study confirmed the usefulness of tocilizumab in corticodependent forms and demonstrated its efficacy. Another IL-6 inhibitor, sarilumab was authorized for the treatment for polymyalgia rheumatic in adult patients with inadequate response to corticosteroid or relapsing disease but is not reimbursed in France.

Baricitinib is an oral selective JAK inhibitor of JAK1 and JAK2 with a short half-life. There are two dosages available (i.e., 2-mg and 4-mg) which can help conduct a simple dose tapering. Administration of baricitinib resulted in a rapid dose dependent inhibition of IL-6 induced STAT3 phosphorylation. An evaluation could be made using the PMR-AS with and without imputation to minimize the effect of baricitinib on CRP by anti-IL-6 effect.

Preliminary results of the BACHELOR study (34 patients treated with baricitinib or placebo) suggested a great efficacy of baricitinib in early PMR without steroids.

It could be a treatment of PMR, with low dose or no steroids only during the first month, to minimize the adverse events of steroids. JAK inhibitors have been reevaluated by EMA, the Oral Surveillance study suggesting that tofacitinib (Xeljanz®) increases the risk of major cardiovascular problems, cancer, VTE, serious infections and death due to any cause when compared with medicines belonging to the class of TNF-alpha inhibitors. EMA has concluded that these safety findings apply to all approved uses of JAK inhibitors in chronic inflammatory disorders. Nevertheless, the risk was not increased during the first months of treatment in all studies and a short treatment could have lower risks than steroids.

As no suitable treatment alternatives are available, excepted GCs which increase the vascular risk and osteoporosis, short treatment by jak inhibitor could be a relevant alternative treatment of PMR. Indeed, the physicians do not have any disease modifying drug (excepted anti IL6 off-label) in treatment of PMR. So, GCs are used for more than one year in the treatment of PMR. Baricitinib, used only 6 months demonstrated its ability to cure early PMR without steroids. It could be an alternative to steroid when physicians consider that ratio benefit/risk is better with a 6 months treatment by baricitininib than >one year by steroids.

Our goal is now to demonstrate in a large cohort the ability of a 6-month treatment with baricitinib in comparison to placebo to decrease glucocorticoids and then to maintain low disease activity without corticosteroids in PMR and a good safety profile.

Due to the possible lower risk of 2 mg than 4 mg of baricitinib, but probably a lower efficacy, the investigators plan to compare both baricitinib (4 mg and 2 mg) to placebo. The study will be conducted in France.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age.
* Fulfilling ACR/EULAR classification criteria for PMR newly diagnosed or treatment resistant.
* No GCs or GCs <15 mg/day since at least 15 days prior to planned randomization.
* PMR-AS-CRP >17.
* Absence of other inflammatory arthropathy, connective tissue diseases or vasculitis.
* Able to give informed consent.
* French health insurance holder

Exclusion Criteria:

* Clinical evidence of giant cell arteritis.
* Uncontrolled high blood pressure or cardiovascular disease.
* High risk of VTE because of a history of VTE (DVT and/or PE) within 12 weeks prior to randomization or a history of recurrent (>1) VTE (counting co-occurring DVT+PE as 1 single event).
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to PMR
* Planned major surgical procedure during the study or medical history, blood abnormalities or any clinical condition that compromises inclusion.
* Current smoker if age >65 years.
* Current active uncontrolled infection.
* Treatment by probenecid.
* Alkaline phosphatase (ALP) ≥2 x ULN.
* Total bilirubin level (TBL) ≥1.5 x ULN.
* Neutropenia (absolute neutrophil count <1000 cells/uL) (<1.00 x 103/uL or <1.00 GI/L).
* Lymphopenia (lymphocyte count <500 cells/uL) (<0.50 x 103/uL or <0.50 GI/L).
* Patient under court protection or protected adults

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2028-11-12 (Estimated); Study Completion 2029-06-12 (Estimated)

PRIMARY OUTCOMES:
Following of the Polymyalgia Rheumatica Activity score | From week 0 to week 24
  Polymyalgia Rheumatica Activity Score (PMR-AS) ≤10 (no flare) without steroids at week 24.
  The Polymyalgia Rheumatica Activity Score is calculated by combining several parameters (patient's pain assessment (using a visual analogue scale) + physician's global assessment of the disease (using a visual analogue scale)+ morning stiffness + C-Reactive Protein level).
  If PMR-AS ≤ 1,5 means remission of the disease. If PMR-AS < 7 means inactive activity of the disease. If 7 <PMR-AS < 17 means low activity of the disease. If PMR-AS > 17 means high activity of the disease.

SECONDARY OUTCOMES:
Following of the Polymyalgia Rheumatica Activity score | From week 0 to week 12
  Polymyalgia Rheumatica Activity score ≤10 (no flare) without steroids at week 12.
  The Polymyalgia Rheumatica Activity Score is calculated by combining several parameters (patient's pain assessment (using a visual analogue scale) + physician's global assessment of the disease (using a visual analogue scale)+ morning stiffness + C-Reactive Protein level).
  If PMR-AS ≤ 1,5 means remission of the disease. If PMR-AS < 7 means inactive activity of the disease. If 7 <PMR-AS < 17 means low activity of the disease. If PMR-AS > 17 means high activity of the disease.
Following of the Polymyalgia Rheumatica Activity score | From week 0 to week 36
  Polymyalgia Rheumatica Activity score ≤10 (no flare) without steroids at week 36.
  The Polymyalgia Rheumatica Activity Score is calculated by combining several parameters (patient's pain assessment (using a visual analogue scale) + physician's global assessment of the disease (using a visual analogue scale)+ morning stiffness + C-Reactive Protein level).
  If PMR-AS ≤ 1,5 means remission of the disease. If PMR-AS < 7 means inactive activity of the disease. If 7 <PMR-AS < 17 means low activity of the disease. If PMR-AS > 17 means high activity of the disease.
Following of the Polymyalgia Rheumatica Activity score | From week 0 to week 36
  Absence of flare according to the investigator at week 36.

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - VIDAL François, Aix-en-Provence
  - LEGRAND Jean-Louis, Arras
  - Besançon-CIC, Besançon
  - PRATI Clément, Besançon
  - CHU de Bordeaux Pellegrin, Bordeaux
  - Dr Alain SARAUX, Brest
  - RAT Anne-Christine, Caen
  - LESKE Charles, Cholet
  - TOURNADRE Anne, Clermont-Ferrand
  - RAMON André, Dijon
  - APHP - Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - DIREZ Guillaume, Le Mans
  - FLIPO René-Marc, Lille
  - WIRTH Théo, Marseille
  - LE HENAFF Catherine, Morlaix
  - CHU de Nice, Nice
  - FAUTREL Bruno - AP-HP La Pitié-Salpétrière, Paris
  - OTTAVIANI Sébastien - AP-HP Bichat, Paris
  - CHU Reims, Reims
  - GOTTENBERG Jacques-Eric, Strasbourg
  - CHU de Toulouse, Toulouse
  - CARVAJAL ALEGRIA Guillermo, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.